CLINICAL TRIAL: NCT04078672
Title: Retinal Imaging Using NOTAL-OCT V3.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NOTAL-OCT V3.0
Record Dates: First submitted 2019-08-27; First posted 2019-09-06 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-04

CONDITIONS: AMD; DR

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMD (Experimental): NOTAL-OCT V3.0 scan
  Interventions: Procedure: NOTAL-OCT V3.0

INTERVENTIONS:
Procedure: NOTAL-OCT V3.0 — AMD and DR patients
  Other Names: OCT scan

SUMMARY:
The study will include up to 250 AMD patients and up to 30 DR patients. In Tel Aviv medical center up to 100 AMD/ 20 DR patients will be recruited; In Assuta HaShalom up to 100 AMD/10 DR patients will be recruited; In Bnei Zion medical center up to 50 AMD patients will be recruited.

4.1 Study population 1. AMD patients - intermediate and advanced AMD (with active or non-active CNV) 2. DR patients - with and without edema 4.2 Inclusion criteria

1. Ability and agreement to give informed consent (IC)
2. Diagnosis of AMD or DR in SE by OCT
3. Ability to undergo OCT scans
4. VA of 20/400 (6/120) or better in study eye(s)

4.3 Exclusion criteria

1. Patient with dilated eye(s)

DETAILED DESCRIPTION:
4.5.1 SCREENING VISIT:

For patients eligible to participate in the study, the following procedure will be done in the screening visit:

1. Patient will sign the IC (Informed Consent) form
2. Test the eligible eye(s) of the patient will be tested
3. The following demographic and clinical data will be collected for each tested eye and will be registered in the CRF:

   1. Patient's DOB and gender.
   2. Patient's diagnosis in study eye(s), based on patient's medical record, including media opacity (e.g. cataract or corneal opacity, if exists).
   3. Examination to check habitual correction, pinhole VA and refraction.

   4.5.2 OCT Visit 1: may take place on the same day as screening visit.

   For each eligible eye, testing will include:

   d. Refraction by auto-refractometer e. Commercial OCT scanning: i. Scanning pattern: Macular cube of at least 6mm (20 degrees); At least 40 B-scans per cube f. NOTAL-OCT V3.0 scanning: i. Scanning pattern Macular cube of the central 10 degrees of the macula At least 40 B-scans per cube ii. The patients will undergo an interactive tutorial that will teach the patient to self-operate the NOTAL-OCT V3.0 device. The tutorial will be done only once, using the eye with the better VA.

   iii. To check repeatability, image capturing phase will include up to 8 testing sessions, each ~2 minutes long.

   iv. Patients will rest for 5 minutes between sessions. v. Total examination time with NOTAL-OCT V3.0 is expected to be less than an hour.

   vi. In case of patient's fatigue during the testing procedure, examination session will be terminated.

   vii. The study staff will administer the NOTAL-OCT V3.0 "patient-experience" questionnaire at the 1st OCT Visit.

   4.5.3 OCT Visits 2-6:

   For each eligible eye, imaging will include:

   a. Commercial OCT scanning: i. Scanning pattern: Macular cube of at least 6mm (20 degrees); At least 40 B-scans per cube b. NOTAL-OCT V3.0 scanning: i. Scanning pattern Macular cube of the central 10 degrees of the macula At least 40 B-scans per cube ii. Image capturing phase that will include up to 8 testing sessions, each a~2 minutes long.

   iii. Patients will rest for 5 minutes between sessions. iv. Total examination time with the NOTAL-OCT V3.0 is expected to be less than an hour.

   v. In case of patient's fatigue during the testing procedure, examination will be terminated.

   c. VA of eye(s) participating in the study. d. Clinical diagnosis of eye(s) participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability and agreement to give informed consent (IC) 2. Diagnosis of AMD or DR in SE by OCT 3. Ability to undergo OCT scans 4. VA of 20/400 (6/120) or better in study eye(s)

Exclusion Criteria:

* 1. Patient with dilated eye(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the level of agreement between OCT images captured by NOTAL-OCT V3.0 and by a commercial OCT | Less then an hour
  The measurement of fluid as identified by an eye-care professional, in the central 10 degrees of the macula of DR patients.

SECONDARY OUTCOMES:
To evaluate the level of agreement between OCT images captured by NOTAL-OCT V3.0 and a by commercial OCT | Less then an hour
  The measurement of fluid as identified by an eye-care professional, in the central 10 degrees of the macula of DR patients.
To evaluate repeatability | Less then an hour
  To evaluate the repeatability of the detection of fluid in images captured by NOTAL-OCT V3.0 in the central 10 degrees of the macula of AMD and DR patients.
To evaluate the level of agreement between NOTAL-OCT V3.0 and a commercial OCT in the presence of fluid | Less then an hour
  The measurement of fluid as identified by an eye-care professional, in the central 10 degrees of the macula.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Assuta Hashalom, Tel Aviv
  - Tel Aviv Medical Center, Tel Aviv